CLINICAL TRIAL: NCT01287793
Title: Randomized, 4-Way, Crossover Single Dose, Placebo And Active Controlled Study To Evaluate The Effect Of Single Intravenous Doses Of Tigecycline On QTc Intervals In Healthy Subjects
Brief Title: Study To Evaluate The Effect Of Single Intravenous Doses Of Tigecycline On QTc Intervals In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1811062
Record Dates: First submitted 2011-01-21; First posted 2011-02-01 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
MeSH Terms: interventions — Tigecycline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- high dose tigecycline (Experimental)
  Interventions: Drug: tigecycline
- regular dose tigecycline (Experimental)
  Interventions: Drug: tigecycline
- moxifloxacin (Active Comparator)
  Interventions: Drug: moxifloxacin; Drug: 100 mL 0.9% Sodium Chloride intravenous
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tigecycline — intravenous, 200 mg, single dose
  Other Names: Tygacil, GAR-936
  Arms: high dose tigecycline
Drug: tigecycline — intravenous, 50 mg, single dose
  Other Names: Tygacil, GAR-936
  Arms: regular dose tigecycline
Drug: moxifloxacin — oral tablet, 400 mg, single dose
  Arms: moxifloxacin
Drug: 100 mL 0.9% Sodium Chloride intravenous — intravenous fluid, 100 mL, single dose
  Arms: moxifloxacin
Drug: placebo — 0.9% Sodium Chloride intravenous 100mL, single dose
  Arms: placebo

SUMMARY:
Administration of a single 50 mg or 200 mg dose of tigecycline will not cause a change in QT/QTc intervals.

DETAILED DESCRIPTION:
evaluation of effect of tigecycline on QT/QTc in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body mass index 17.5 - 30.5 kg
* Total body weight greater than 50 kg

Exclusion Criteria:

* Recent history of diarrhea
* Use of oral antibiotics in the last 2 weeks
* History of risk factors for QT prolongation pregnant females
* Nursing females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serial QTc measurements in healthy volunteers up to 96 hours after single tigecycline doses | Up to 96 hours

SECONDARY OUTCOMES:
QTc, using Fredericia's correction at each time point during moxifloxacin treatment periods | -2.5, -2, -1.5, -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Maximum concentration pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Time of maximum concentration pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Elimination rate constant pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Half life pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Area under the concentration time curve to last measured concentrations pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Area under the concentration time curve extrapolated to infinity pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Clearance pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Volume of distribution at steady-state pharmacokinetic endpoint for tigecycline | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours
Response-exposure relationships between QT/QTc and tigecycline concentration | -1, 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Korth-Bradley JM, McGovern PC, Salageanu J, Matschke K, Plotka A, Pawlak S. Tigecycline does not prolong corrected QT intervals in healthy subjects. Antimicrob Agents Chemother. 2013 Apr;57(4):1895-901. doi: 10.1128/AAC.01576-12. Epub 2013 Feb 12. PMID 23403419
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1811062&StudyName=Study%20To%20Evaluate%20The%20Effect%20Of%20Single%20Intravenous%20Doses%20Of%20Tigecycline%20On%20QTc%20Intervals%20In%20Healthy%20Subjects